CLINICAL TRIAL: NCT07056621
Title: Does Belimumab Modify the Natural History of SLE? A Propensity Score-matched, Real-world Study
Status: Recruiting | Type: Observational
Sponsor: Biomedical Research Foundation, Academy of Athens (Other)
Responsible Party: Principal Investigator, DIMITRIOS BOUMPAS, Professor in Medicine, Biomedical Research Foundation, Academy of Athens
Other Study IDs: 224080
Record Dates: First submitted 2025-06-30; First posted 2025-07-09 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-06

CONDITIONS: SLE - Systemic Lupus Erythematosus
Keywords: SLE; belimumab; bilag
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group A: Belimumab: Group A will consist of patients under treatment with belimumab.
- Group B: Standard-of-care (follow-up after May 1st 2014): Group B will consist of patients on standar-of-care SLE treatment, who were followed-up after May 1st 2014 (the first date where belimumab was available in Greece).
- Group C: Standar-of-care (follow-up before May 1st 2014): Group C will consist of a historical cohort of patients under standar-of-care, followed-up before May 1st 2014 (the first date where belimumab was available in Greece).

SUMMARY:
This will be a combined retrospective and prospective cohort study, that will evaluate the incidence of de novo Systemic Lupus Erythematosus major organ manifestations (defined as BILAG A flares) in patients receiving belimumab (Arm A) and compare it to 2 standard-of-care groups (SoC) (Arm B: patients on SoC; Arm C: patients on SoC followed-up up to May 1st 2014, the first date where belimumab was available in Greece).

The investigators will utilize survival analysis methods (Kaplan-Meier survival curves and Cox regression) and mixed effects longitudinal analyses. Additionally, the investigators will employ propensity score matching and/or inverse probability of treatment weighting, to create balanced cohorts and reduce bias.

DETAILED DESCRIPTION:
Belimumab (BEL) has been used for the treatment of SLE for over 10 years, with clear evidence for a beneficial effect in reduction of disease activity and frequency of flares, as well as prevention of damage accrual.

Whether BEL may also result in prevention of incident, major organ involvement in patients with SLE is less clear. A recent post-hoc analysis of the BLISS trials suggested that BEL (although at the low, rather than standard-dose) reduced the rate of de novo renal flares (defined by BILAG) compared to standard-of-care but real-life data are scarce. Importantly, data on the ability of belimumab to decrease major neuropsychiatric events in SLE such as strokes, seizures and cognitive dysfunction or other severe manifestations such as severe hematologic or cardiopulmonary disease is not known.

To this end, the investigators propose a propensity score-matched, real-world, with the use of longitudinal data from large patient cohorts and time-to-event analyses. Given the non-experimental setting of this study, the investigators will also employ propensity score matching (PSM), to create balanced cohorts of BEL-treated and non-BEL-treated patients and reduce bias in estimating treatment efficacy.

The study will consist of 3 arms, as follows: Arm A: patients on treatment with belimumab; Arm B: patients on standard-of-care (SoC) treatment from May 1st 2014 onwards; Arm C: a historical cohort of patients on SoC followed-up up to May 1st 2014, the first date where belimumab was available in Greece.

ELIGIBILITY:
Inclusion Criteria:

* Systemic lupus erythematosus classification according to the Systemic Lupus International Collaborating Clinics (SLICC) criteria
* Age ≥ 18 years old
* Time of follow-up ≥ 6 months
* Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) ≥ 4
* Physician Global Assessment (PGA) visual analogue score > 1

Exclusion Criteria:

* Patients with incomplete medical records or missing key variables
* Patients with concomitant autoimmune disorders (excluding thyroid disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult systemic lupus erythematosus patients, receiving belimumab (Arm A) or standard-of-care treatment (Arms B and C).
Sampling Method: Probability Sample
Enrollment: 684 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Bilag A flare | From enrollment to the end of treatment (expected follow-up duration 1-4 years).
  Major organ systemic lupus erythematosus manifestations as defined by the BILAG (British Isles Lupus Assessment Group) index (BILAG A flare)

SECONDARY OUTCOMES:
SLICC/ACR Damage Index | From enrollment to the end of treatment (expected follow-up duration 1-4 years).
  Systemic Lupus International Collaborating Clinics, ACR/American College of Rheumatology (SLICC/ACR) Damage Index (SDI)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital 'Attikon', Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No
The investigators are not currently planning on sharing Individual participant data (IPD). This decision is based on the fact the investigators have not made specific agreements with our hospital's IRB about individual participant data sharing. Study results will be disseminated through peer-reviewed publications, which will provide comprehensive findings while maintaining participant confidentiality. However, upon reasonable requests from qualified researchers for legitimate scientific purposes, the investigators may consider sharing de-identified IPD on a case-by-case basis, after approval by our IRB.

REFERENCES:
- [Background] Fanouriakis A, Adamichou C, Koutsoviti S, Panopoulos S, Staveri C, Klagou A, Tsalapaki C, Pantazi L, Konsta S, Mavragani CP, Dimopoulou D, Ntali S, Katsikas G, Boki KA, Vassilopoulos D, Konstantopoulou P, Liossis SN, Elezoglou A, Tektonidou M, Sidiropoulos P, Erden A, Sfikakis PP, Bertsias G, Boumpas DT. Low disease activity-irrespective of serologic status at baseline-associated with reduction of corticosteroid dose and number of flares in patients with systemic lupus erythematosus treated with belimumab: A real-life observational study. Semin Arthritis Rheum. 2018 Dec;48(3):467-474. doi: 10.1016/j.semarthrit.2018.02.014. Epub 2018 Feb 23. PMID 29555348
- [Background] Nikoloudaki M, Nikolopoulos D, Koutsoviti S, Flouri I, Kapsala N, Repa A, Katsimbri P, Theotikos E, Pitsigavdaki S, Pateromichelaki K, Bertsias A, Elezoglou A, Sidiropoulos P, Fanouriakis A, Boumpas D, Bertsias G. Clinical response trajectories and drug persistence in systemic lupus erythematosus patients on belimumab treatment: A real-life, multicentre observational study. Front Immunol. 2023 Jan 4;13:1074044. doi: 10.3389/fimmu.2022.1074044. eCollection 2022. PMID 36685524
- [Background] Iaccarino L, Bettio S, Reggia R, Zen M, Frassi M, Andreoli L, Gatto M, Piantoni S, Nalotto L, Franceschini F, Larosa M, Fredi M, Punzi L, Tincani A, Doria A. Effects of Belimumab on Flare Rate and Expected Damage Progression in Patients With Active Systemic Lupus Erythematosus. Arthritis Care Res (Hoboken). 2017 Jan;69(1):115-123. doi: 10.1002/acr.22971. Epub 2016 Nov 18. PMID 27390293
- [Background] Bartels C, Bell C, Rosenthal A, Shinki K, Bridges A. Decline in rheumatoid vasculitis prevalence among US veterans: a retrospective cross-sectional study. Arthritis Rheum. 2009 Sep;60(9):2553-7. doi: 10.1002/art.24775. PMID 19714622
- [Background] van Vollenhoven R, Askanase AD, Bomback AS, Bruce IN, Carroll A, Dall'Era M, Daniels M, Levy RA, Schwarting A, Quasny HA, Urowitz MB, Zhao MH, Furie R. Conceptual framework for defining disease modification in systemic lupus erythematosus: a call for formal criteria. Lupus Sci Med. 2022 Mar;9(1):e000634. doi: 10.1136/lupus-2021-000634. PMID 35346982
- [Background] Fanouriakis A, Kostopoulou M, Andersen J, Aringer M, Arnaud L, Bae SC, Boletis J, Bruce IN, Cervera R, Doria A, Dorner T, Furie RA, Gladman DD, Houssiau FA, Ines LS, Jayne D, Kouloumas M, Kovacs L, Mok CC, Morand EF, Moroni G, Mosca M, Mucke J, Mukhtyar CB, Nagy G, Navarra S, Parodis I, Pego-Reigosa JM, Petri M, Pons-Estel BA, Schneider M, Smolen JS, Svenungsson E, Tanaka Y, Tektonidou MG, Teng YO, Tincani A, Vital EM, van Vollenhoven RF, Wincup C, Bertsias G, Boumpas DT. EULAR recommendations for the management of systemic lupus erythematosus: 2023 update. Ann Rheum Dis. 2024 Jan 2;83(1):15-29. doi: 10.1136/ard-2023-224762. PMID 37827694